CLINICAL TRIAL: NCT04779411
Title: Validation of a Lutein and Zeaxanthin Food Frequency Questionnaire, and an Electronic Device Use Questionnaire.
Brief Title: Online Validation of Dietary Intake Food Frequency Questionnaire Over Four Weeks, and Electronic Device Use Questionnaire Over Eight Weeks.
Status: Completed | Type: Observational
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Other Study IDs: FFQEDUQ20V1
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2022-05

CONDITIONS: Lutein and Zeaxanthin Dietary Intake; Age Related Macular Degeneration; Blue Light Exposure; Electronic Device Use
Keywords: Lutein; Zeaxanthin; Food Frequency Questionnaire; Blue Light; Electronic Device Use
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Food Frequency Questionnaire Validation Group: The validation procedure will span over four weeks, consisting of administering the Lutein and Zeaxanthin Food Frequency Questionnaire (FFQ L/Z) and 24-hour diet recalls at multiple timepoints. Timepoints for the eight 24-hour diet recalls will be determined by random number generator for each of the participants at baseline (https://www.random.org/), of which two will take place on weekend days, and the remainder on week days.
  * The weekly L/Z FFQ will be completed at the conclusion of each of the four weeks.
  * The monthly L/Z FFQ will be completed at baseline and at the conclusion of week four.
  Interventions: Other: Weekly Food Frequency Questionnaire; Other: Monthly Food Frequency Questionnaire; Other: 24-Hour Diet Recall
- Electronic Device Use Questionnaire Validation Group: The validation procedure will occur over eight weeks consisting of administering eight 24-hour diary of electronic device use (24-hour ED use diary) and the Electronic Device Use Questionnaire (EDUQ) at three time points. The time points for the eight 24-hour ED use diaries will be determined by random number generator for each of the participants at baseline (https://www.random.org/), of which two will take place on weekend days, and the remainder on weekdays. The EDUQ will be completed at baseline and at the conclusion of weeks four and eight.
  Interventions: Other: Electronic Device Use Questionnaire; Other: 24-Hour Electronic Device Use Diary

INTERVENTIONS:
Other: Weekly Food Frequency Questionnaire — A purpose designed 91-item questionnaire to measure frequency of consumption of a selection of L/Z containing foods over the prior 7 days.
  Groups: Food Frequency Questionnaire Validation Group
Other: Monthly Food Frequency Questionnaire — A purpose designed 95-item questionnaire completed at visit 1 to measure frequency of consumption of a selection of L/Z containing foods over the prior month.
  Groups: Food Frequency Questionnaire Validation Group
Other: 24-Hour Diet Recall — the diet recall via the online Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24®) takes approximately 25 minutes to complete, and investigates food and beverages consumed in the prior 24-hours.
  Groups: Food Frequency Questionnaire Validation Group
Other: Electronic Device Use Questionnaire — 1. The EDUQ: A 22-item questionnaire that takes 20 minutes to complete, and measures participant demographic information (weight, height, age, highest level of education, occupational status, post-code and country of residence), usual daily ED use from present up to 20 years ago, occupational influence to use, and differences to ED use between a weekend and weekday.
  Groups: Electronic Device Use Questionnaire Validation Group
Other: 24-Hour Electronic Device Use Diary — Participants asked to record their electronic device use in hours and minutes over 24 hours.
  Groups: Electronic Device Use Questionnaire Validation Group

SUMMARY:
Tools to investigate dietary lutein and zeaxanthin (L/Z) intake and electronic device (ED) use are important to progress research that investigates the role of ED blue light (BL) exposure, and dietary L/Z intake on macular health. This project aims to validate two questionnaires developed by our research group: The L/Z FFQ, and the Electronic Device Use Questionnaire (EDUQ). The L/Z FFQ aims to investigate dietary intake of L/Z over the prior week or month. The EDUQ aims to investigate usual hours and behaviours surrounding ED use over the prior three months.

This aims of this project are to:

1. Validate a L/Z FFQ recalling over a weekly and monthly timeframe against multiple 24-hour diet recalls over four weeks.
2. Validate the EDUQ against multiple 24-hour ED use diaries over eight weeks. A cohort of 100 adults will be invited to participate to validate the FFQ and EDUQ. Participants will be offered to choose to participate in one or both the questionnaire validations (L/Z FFQ and EDUQ).

DETAILED DESCRIPTION:
L/Z FFQ Validation The validation procedure will span over four weeks, consisting of administering the L/Z FFQ and 24-hour diet recalls at multiple timepoints. Timepoints for the eight 24-hour diet recalls will be determined by random number generator for each of the participants at baseline (https://www.random.org/), of which two will take place on weekend days, and the remainder on week days.

* The weekly L/Z FFQ will be completed at the conclusion of each of the four weeks.
* The monthly L/Z FFQ will be completed at baseline and at the conclusion of week four.

Participants will indicate their consent to participate on Checkbox® by proceeding to the complete the questionnaires.

1. Demographic information: at the beginning of the first investigation (monthly L/Z FFQ) participants will be asked to report their weight, height, age, gender, highest level of education, occupational status (employed or unemployed), post-code and country of residence, usual hours of physical activity per week, how they heard about the study, and whether they are actively trying to gain or lose weight. Personal information is to be collected to qualify the characteristics of the population in which the tool is being validated. Data collected via Checkbox ®.
2. L/Z FFQ: The weekly L/Z FFQ is a 91-item questionnaire that takes approximately 20 minutes to complete, and investigates the frequency of intake of listed foods or supplements over the prior seven days. The monthly L/Z FFQ contains the same 91 items, takes approximately 30 minutes to complete, and investigates the frequency of intake of listed foods or supplements over the prior month. In addition, the monthly L/Z FFQ contains four qualitative questions that investigate change in usual dietary intake over the last one to ten years. Questionnaire data collected via Checkbox®.
3. 24-hour diet recall: the diet recall via the online Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24®) takes approximately 25 minutes to complete, and investigates food and beverages consumed in the prior 24-hours (20). The ASA24® is supported by the National Institutes of Health (NIH) in the United States (US) with national variants and as a US government entity not within the EU-US Data Privacy Shield for legal reasons. Therefore, explicit consent for use of the ASA24® tool will be sought from participants. For further information on the tool: https://epi.grants.cancer.gov/asa24/.

EDUQ Validation

The validation procedure will occur over eight weeks consisting of administering eight 24-hour diary of ED use (24-hour ED use diary) and the EDUQ at three time points. The time points for the eight 24-hour ED use diaries will be determined by random number generator for each of the participants at baseline (https://www.random.org/), of which two will take place on weekend days, and the remainder on weekdays. The EDUQ will be completed at baseline and at the conclusion of weeks four and eight. Upon consenting to participate on the Checkbox® by proceeding to the questionnaires, participants will be instructed to fill out:

1. The EDUQ: A 22-item questionnaire that takes 20 minutes to complete, and measures participant demographic information (weight, height, age, highest level of education, occupational status, post-code and country of residence), usual daily ED use from present up to 20 years ago, occupational influence to use, and differences to ED use between a weekend and weekday (questionnaire adapted from Williams et al. (2019) (21). Personal information collected as part of this questionnaire is to qualify the characteristics of the population in which the tool is being validated. Data collected via Checkbox®.
2. 24-hour ED use diary: Participants will be asked to record their ED use in hours and minutes over 24 hours. Data collected via Checkbox®.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females 18 years and over.
* Access to an ED such as a computer, phone, or tablet, and internet to complete investigations.

Exclusion Criteria:

* Visual, hearing, or physical impairment that may prevent from completing investigations.
* No English literacy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Generally healthy male and female adults from Australia or the United Kingdom.
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Daily Intake of lutein and zeaxanthin | 4 weeks
  Calculation from each dietary intake tool what the daily milligrams of lutein and zeaxanthin intake is.
Daily hours of electronic device use. | 8 weeks
  Calculation from the two device use recording tools what the daily hours of electronic device use is for each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Queensland, Saint Lucia, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keel S, Xie J, Foreman J, van Wijngaarden P, Taylor HR, Dirani M. Prevalence of Age-Related Macular Degeneration in Australia: The Australian National Eye Health Survey. JAMA Ophthalmol. 2017 Nov 1;135(11):1242-1249. doi: 10.1001/jamaophthalmol.2017.4182. PMID 29049463
- [Background] Bernstein PS, Li B, Vachali PP, Gorusupudi A, Shyam R, Henriksen BS, Nolan JM. Lutein, zeaxanthin, and meso-zeaxanthin: The basic and clinical science underlying carotenoid-based nutritional interventions against ocular disease. Prog Retin Eye Res. 2016 Jan;50:34-66. doi: 10.1016/j.preteyeres.2015.10.003. Epub 2015 Nov 2. PMID 26541886
- [Background] Velilla S, Garcia-Medina JJ, Garcia-Layana A, Dolz-Marco R, Pons-Vazquez S, Pinazo-Duran MD, Gomez-Ulla F, Arevalo JF, Diaz-Llopis M, Gallego-Pinazo R. Smoking and age-related macular degeneration: review and update. J Ophthalmol. 2013;2013:895147. doi: 10.1155/2013/895147. Epub 2013 Dec 4. PMID 24368940
- [Background] Chiu CJ, Chang ML, Zhang FF, Li T, Gensler G, Schleicher M, Taylor A. The relationship of major American dietary patterns to age-related macular degeneration. Am J Ophthalmol. 2014 Jul;158(1):118-127.e1. doi: 10.1016/j.ajo.2014.04.016. Epub 2014 Apr 29. PMID 24792100
- [Background] Wu J, Seregard S, Algvere PV. Photochemical damage of the retina. Surv Ophthalmol. 2006 Sep-Oct;51(5):461-81. doi: 10.1016/j.survophthal.2006.06.009. PMID 16950247
- [Background] Algvere PV, Marshall J, Seregard S. Age-related maculopathy and the impact of blue light hazard. Acta Ophthalmol Scand. 2006 Feb;84(1):4-15. doi: 10.1111/j.1600-0420.2005.00627.x. PMID 16445433
- [Background] Behar-Cohen F, Martinsons C, Vienot F, Zissis G, Barlier-Salsi A, Cesarini JP, Enouf O, Garcia M, Picaud S, Attia D. Light-emitting diodes (LED) for domestic lighting: any risks for the eye? Prog Retin Eye Res. 2011 Jul;30(4):239-57. doi: 10.1016/j.preteyeres.2011.04.002. Epub 2011 May 14. PMID 21600300
- [Background] Widomska J, Subczynski WK. Why has Nature Chosen Lutein and Zeaxanthin to Protect the Retina? J Clin Exp Ophthalmol. 2014 Feb 21;5(1):326. doi: 10.4172/2155-9570.1000326. PMID 24883226
- [Background] Liu T, Liu WH, Zhao JS, Meng FZ, Wang H. Lutein protects against beta-amyloid peptide-induced oxidative stress in cerebrovascular endothelial cells through modulation of Nrf-2 and NF-kappab. Cell Biol Toxicol. 2017 Feb;33(1):57-67. doi: 10.1007/s10565-016-9360-y. Epub 2016 Nov 22. PMID 27878403
- [Background] Frede K, Ebert F, Kipp AP, Schwerdtle T, Baldermann S. Lutein Activates the Transcription Factor Nrf2 in Human Retinal Pigment Epithelial Cells. J Agric Food Chem. 2017 Jul 26;65(29):5944-5952. doi: 10.1021/acs.jafc.7b01929. Epub 2017 Jul 13. PMID 28665123
- [Background] Satia JA, Watters JL, Galanko JA. Validation of an antioxidant nutrient questionnaire in whites and African Americans. J Am Diet Assoc. 2009 Mar;109(3):502-8, 508.e1-6. doi: 10.1016/j.jada.2008.11.033. PMID 19248870
- [Background] Romieu I, Parra S, Hernandez JF, Madrigal H, Willett W, Hernandez M. Questionnaire assessment of antioxidants and retinol intakes in Mexican women. Arch Med Res. 1999 May-Jun;30(3):224-39. doi: 10.1016/s0188-0128(99)00017-2. PMID 10427874
- [Background] McNaughton SA, Marks GC, Gaffney P, Williams G, Green A. Validation of a food-frequency questionnaire assessment of carotenoid and vitamin E intake using weighed food records and plasma biomarkers: the method of triads model. Eur J Clin Nutr. 2005 Feb;59(2):211-8. doi: 10.1038/sj.ejcn.1602060. PMID 15483635
- [Background] Stringham JM, Stringham NT, O'Brien KJ. Macular Carotenoid Supplementation Improves Visual Performance, Sleep Quality, and Adverse Physical Symptoms in Those with High Screen Time Exposure. Foods. 2017 Jun 29;6(7):47. doi: 10.3390/foods6070047. PMID 28661438
- [Background] Cartmel B, Moon TE. Comparison of two physical activity questionnaires, with a diary, for assessing physical activity in an elderly population. J Clin Epidemiol. 1992 Aug;45(8):877-83. doi: 10.1016/0895-4356(92)90071-t. PMID 1624970
- [Background] Park Y, Dodd KW, Kipnis V, Thompson FE, Potischman N, Schoeller DA, Baer DJ, Midthune D, Troiano RP, Bowles H, Subar AF. Comparison of self-reported dietary intakes from the Automated Self-Administered 24-h recall, 4-d food records, and food-frequency questionnaires against recovery biomarkers. Am J Clin Nutr. 2018 Jan 1;107(1):80-93. doi: 10.1093/ajcn/nqx002. PMID 29381789
- [Background] Williams R, Bakshi S, Ostrin EJ, Ostrin LA. Continuous Objective Assessment of Near Work. Sci Rep. 2019 May 6;9(1):6901. doi: 10.1038/s41598-019-43408-y. PMID 31061427
- [Background] Black AE. Critical evaluation of energy intake using the Goldberg cut-off for energy intake:basal metabolic rate. A practical guide to its calculation, use and limitations. Int J Obes Relat Metab Disord. 2000 Sep;24(9):1119-30. doi: 10.1038/sj.ijo.0801376. PMID 11033980
- [Background] Black AE. The sensitivity and specificity of the Goldberg cut-off for EI:BMR for identifying diet reports of poor validity. Eur J Clin Nutr. 2000 May;54(5):395-404. doi: 10.1038/sj.ejcn.1600971. PMID 10822286
- See also: USDA Food Composition Database — https://fdc.nal.usda.gov/